CLINICAL TRIAL: NCT06185166
Title: State of Play of Non-tuberculous Mycobacteria in Alsace: a Retrospective Study
Brief Title: State of Play of Non-tuberculous Mycobacteria in Alsace
Acronym: Mycoba
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: University Hospital, Strasbourg, France (Other)
Responsible Party: Sponsor
Other Study IDs: 8780
Record Dates: First submitted 2023-12-14; First posted 2023-12-29 (Actual); Last update posted 2023-12-29 (Actual); Status verified 2023-12

CONDITIONS: Non-Tuberculous Mycobacteria
Keywords: Non-Tuberculous Mycobacteria

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Non-tuberculous mycobacteriosis (NTM) are infectious diseases caused by mycobacteria that are not part of the Tuberculosis complex. More than 190 species have been identified to date.

As an environmental reservoir, it most often affects the lungs, skin and soft tissues, lymph nodes, but it can affect all organs. Varying in virulence depending on the species, most infections do not cause illness.

There is currently no coordinated care pathway for this pathology in Alsace. The means necessary to set up such a structure requires knowing the importance of the disease.

DETAILED DESCRIPTION:
The aim of the study is to determine the incidence of non-tuberculous mycobacterial infections in the ALSACE region, the proportion of cases in which the infection causes illness, and its evolution over time.

ELIGIBILITY:
Inclusion Criteria:

* Adult subject (≥ 18 years old)
* in whom a biological sample is culture positive for a non-tuberculous mycobacterium
* born in France and domiciled in Alsace (i.e. whose home postal code begins with 67 or 68)
* not opposing the reuse of its data for scientific research purposes

Exclusion Criteria:

* Subject having expressed opposition to participating in the study
* not domiciled in Alsace
* Born abroad
* Isolation of a mycobacterium from the Tuberculosis complex and Mycobacterium gordonae

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Study Population: Adult subject (≥ 18 years old) in whom a biological sample is culture positive for a non-tuberculous mycobacterium
Sampling Method: Non-Probability Sample
Enrollment: 100 (Estimated)
Dates: Start 2022-12-05 (Actual); Primary Completion 2024-06 (Estimated); Study Completion 2024-06-05 (Estimated)

PRIMARY OUTCOMES:
Retrospective description of non-tuberculous mycobacteria in Alsace | Through study completion, an average of 6 months

CONTACTS AND LOCATIONS:
Locations (1):
- Service de Pneumologie - CHU de Strasbourg - France, Strasbourg, France